CLINICAL TRIAL: NCT04128488
Title: Effects of Gender-Affirming Hormone Therapy Among Transgender Women
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH); American Heart Association (Other); Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Mabel Toribio, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2019P001962; 1K23HL147799-01 (NIH)
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Transgender Women; HIV/AIDS; Cardiovascular Diseases; Metabolic Disease; Coagulopathy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases; Metabolic Diseases; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transgender women and non-binary individuals without HIV
  Interventions: Other: Abdominal MR Imaging; Other: Cardiac MRI/MRS; Other: Oral Glucose Tolerance Testing; Other: Whole Body, Lumbar Spine, and Hip DEXA Imaging
- Transgender women and non-binary individuals with HIV
  Interventions: Other: Abdominal MR Imaging; Other: Cardiac MRI/MRS; Other: Oral Glucose Tolerance Testing; Other: Whole Body, Lumbar Spine, and Hip DEXA Imaging

INTERVENTIONS:
Other: Abdominal MR Imaging — Imaging to evaluate visceral adipose tissue and hepatic lipid content
Other: Cardiac MRI/MRS — Imaging to evaluate cardiac function and structure
Other: Oral Glucose Tolerance Testing — Blood testing to evaluate changes in glucose and insulin in response to oral glucose load
Other: Whole Body, Lumbar Spine, and Hip DEXA Imaging — Imaging to evaluate fat and lean body mass as well as bone mineral density

SUMMARY:
In this study, investigators plan to evaluate the cardiometabolic effects of initiating gender-affirming hormone therapy among transgender women with and without HIV. As part of this study, participants will undergo cardiovascular and metabolic phenotyping within 3 months of starting and after 12 months of gender-affirming hormone therapy. Cardiovascular phenotyping will include cardiac MRI/MRS imaging to evaluate cardiac function and structure. Metabolic phenotyping will include oral glucose tolerance testing, abdominal MR imaging to evaluate visceral adiposity, and whole body, lumbar, and hip DEXA imaging to evaluate fat and lean body mass as well as bone mineral density, respectively. Traditional markers of CVD risk as well as immune, hormonal, and coagulation parameters will also be assessed longitudinally.

ELIGIBILITY:
Inclusion Criteria:

* transgender women or non-binary individual
* age ≥16
* For women with HIV only: on ART therapy for ≥3 months
* initiation of testosterone suppression with spironolactone or leuprolide and estrogen therapy with oral 17-β estradiol, transdermal 17β estradiol, sublingual estradiol, intramuscular estradiol, or subcutaneous estradiol by medical provider

Exclusion Criteria:

* For women with HIV only: CD4 count<50
* history of CAD, ACS, ASCVD risk score ≥ 7.5%, LDL-C ≥ 190, or angina (e.g. current indication for statin use)
* history of heart failure
* history of diabetes
* eGFR < 30 ml/min/1.73m2
* standard contraindication to MRI, including history of severe allergy to gadolinium or Dotarem
* prior orchiectomy
* gender-affirming hormone therapy for greater than 5 months directly prior to enrollment
* current or past anti-platelet therapy or anti-coagulant therapy within the last 6 months •current or past statin therapy within the last 6 months
* concurrent enrollment in conflicting research study

Ages: 16 Years to 99 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Transgender Women
Study Population: Transgender Women and Non-Binary Individuals
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Change in Visceral Adipose Tissue | Baseline and 12 months

SECONDARY OUTCOMES:
Change in Intramyocardial Triglyceride Content on Cardiac MRS | Baseline and 12 months
Change in Diastolic Function on Cardiac MRI | Baseline and 12 months
Change in Myocardial Fibrosis on Cardiac MRI | Baseline and 12 months
Change in Glucose and Insulin Parameters on Oral Glucose Tolerance Testing | Baseline and 12 months
Change in Bone Density | Baseline and 12 months
Change in Hormonal Parameters | Baseline and 12 months
Change in Coagulation Parameters | Baseline and 12 months
Change in hepatic lipid content | Baseline and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Talathi R, Juhasz V, Delgado M, Quinaglia T, Ghamari A, Wang M, Alhallak I, Stinebaugh S, Campbell S, Stockman SL, Ozturk MA, Ahmadi SM, Looby SE, Lee H, Poteat TC, Szczepaniak LS, Zanni MV, Neilan TG, Toribio M. Visceral adipose tissue and liver fat on 17-beta estradiol-dominant gender-affirming hormone therapy: A US-based cohort. J Clin Endocrinol Metab. 2025 Dec 12:dgaf665. doi: 10.1210/clinem/dgaf665. Online ahead of print. PMID 41383103